CLINICAL TRIAL: NCT00133562
Title: Prospective Double Blind Randomized Clinical Trial of Alanyl-Glutamine or Glycine in Hospitalized Children With Persistent Diarrhea or Malnutrition.
Brief Title: HIAS II - Study of Nutritional Supplementation in Hospitalized Children With Persistent Diarrhea or Malnutrition
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Richard Guerrant, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11375
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2008-10-28 (Estimated); Status verified 2008-10

CONDITIONS: Diarrhea, Malnutrition; Other Nutritional Deficiencies
Keywords: Malnutrition, pediatric, Brazil, alanyl-glutamine
MeSH Terms: conditions — Diarrhea; Malnutrition | interventions — alanylglutamine; Glycine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alanyl-glutamine
Drug: Glycine

SUMMARY:
This study will determine the effect of 7 days supplementation of alanyl-glutatime or glycine on the damaged intestinal barrier function on day 8 in children with persistent diarrhea or malnutrition.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effect of 7 days supplementation of alanyl-glutamine or glycine on the damaged intestinal barrier function, measured by lactulose/mannitol test on day 8, in children with persistent diarrhea or malnutrition; on diarrhea frequency and duration, weight gain, protein loss, intestinal inflammation, and lactoferrin excretion.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 3 to 36 months with a history of persistent diarrhea (3 or more unformed stools/day) for >2 weeks or height-for-age Z-score (HAZ) less than negative 1, which is the median of HAZ score in children at HIAS.
2. Be an inpatient and willing to stay for 7 nights at HIAS.
3. Child´s parent or guardian must sign informed consent..

Exclusion Criteria:

1. Children exclusively breast-fed (Reason: The diet needs to be controlled in order to evaluate the study treatment effect)
2. Children who participated in the community study or any other study within the past two years (Reason: The children in the community study will have received glutamine.)
3. Children with suspected other illnesses as indicated by fever >102º F at time of screening off antipyretics
4. Children with suspected systemic disease at the time of screening including but not limited to shock, meningitis, sepsis, pneumonia, tuberculosis, varicella
5. Severe malnutrition defined as HAZ <-3 or WAZ <-3.5 or any child weighing <10 lbs. (4.5 kg) or any child with a weight-to-height ratio <60% of the NCHS age adjusted norm.

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108
Dates: Start 2004-08; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Guerrant, MD, Principal Investigator — University of Virginia